CLINICAL TRIAL: NCT01988844
Title: Manual Dexterity and Upper Limbs Functionality Assessment in School Children With Cerebral Palsy
Brief Title: Upper Limbs Assessment in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Other Study IDs: DF0042UG
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Cerebral Palsy; Children
Keywords: functionality; Cerebral palsy; Handwriting
MeSH Terms: conditions — Cerebral Palsy | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children with cerebral palsy: Children diagnosed with cerebral palsy are included in this group. An assessment and an intervention will be carried out.
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — The children with cerebral palsy were assessed. Different measures evaluating the upper limbs functionality are used.
  Other Names: Evaluation; Description

SUMMARY:
Cerebral palsy is the leading cause of physical disability among children. Manual dexterity and upper limbs functionality is limited between these children. The purpose of this study is to stablish a specific profile of school children with cerebral palsy based on the upper limbs assessment.

DETAILED DESCRIPTION:
While the rates of perinatal and infant mortality have declined toward the end of the last century,the rate of cerebral palsy has remained at 2 to 2.5 per 1,000 live births. A high percentage of children with cerebral palsy have difficulty keeping up with the handwriting demands at school. The neurological impairments in children with cerebral palsy frequently limit the functionality of these children taken in to account the upper limbs variables. It should be interesting to describe a clinical profile based on this assessment.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy diagnosis.
* Aged between 6 and 10 years old.
* Children attending a school.

Exclusion Criteria:

* Severe cognitive impairment.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: School children with cerebral palsy.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pediatric Evaluation of Disability Inventory (PEDI) | baseline
  This inventory assess the key functional capabilities and performance in children between six months to seven years old. Three subscales are observed: self-care, mobility and social function. It helps you to identify areas of new functional intervention. Also, it is used to identify functional deficits.
Upper limbs functionality | baseline
  The functionality is measured using the Abilhand-kids questionnaire. This questionnaire was designed to cover the widest range of children's manual activities including both unimanual and bimanual activities. For each question, the children and their parents were asked to provide their perceived difficulty to perform the activity on a three-level scale: impossible (0), difficult (1), or easy (2).

SECONDARY OUTCOMES:
Manual dexterity | baseline
  Manual dexterity is measured using the 9-hole peg test. This is a brief, standardized, quantitative test of upper extremity function. Both the dominant and non-dominant hands are tested twice. The patient is seated at a table with a small container holding nine pegs. The patient picks up the nine pegs one at a time as quickly as possible, puts them in the nine holes, and, once they are in the holes, removes them again as quickly as possible one at a time, replacing them into the shallow container. The time is recorded.
Executive function | baseline
  The executive function is measured using the Porteus Maze Test. It consists of a series of mazes graded in difficulty and standardized for application to children from three years old.
Handwriting assessment | baseline
  The handwriting ability is measured with the Handwriting without tears method. It is used to assess memory, letter size,space and movement control.
Range of motion | baseline
  The range of motion in upper limbs is measured with a standard goniometer at different levels: elbow, wrist and fingers.
Upper limbs strength | baseline
  The strength is evaluated using a digital dynamometer. The strength is measured in Newtons.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Spain, Spain

IPD SHARING:
Plan to Share IPD: Undecided